CLINICAL TRIAL: NCT01931618
Title: Digital Therapy: Evaluation of the Fully Automated Alcohol Intervention "Balance".
Brief Title: Testing the Efficacy of an Online Alcohol Intervention in a Workplace Setting
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oslo (Other)
Collaborators: The Research Council of Norway (Other)
Responsible Party: Principal Investigator, Håvar Brendryen, Senior researcher, University of Oslo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: SERAF-BALANCE-2; 142956 (Other Grant/Funding Number: Norwegian Centre for Addiction Research, University of Oslo)
Record Dates: First submitted 2013-08-26; First posted 2013-08-29 (Estimated); Last update posted 2017-09-08 (Actual); Status verified 2017-09

CONDITIONS: Hazardous Drinking; Harmful Drinking
Keywords: alcohol; online intervention; hazardous drinking; harmful drinking; early intervention; behavior change intervention

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Usual care (Active Comparator): Receives two interventions:
  1. Online screening and feedback.
  2. Online booklet.
  Interventions: Behavioral: Online screening and feedback; Behavioral: Online booklet.
- Extended follow-up (Experimental): Receives two interventions:
  1. Online screening and feedback.
  2. Online multi session follow-up.
  Interventions: Behavioral: Online screening and feedback; Behavioral: Online multi session follow-up

INTERVENTIONS:
Behavioral: Online screening and feedback — An online single session screening procedure including individualized normative feedback.
Behavioral: Online booklet. — An online booklet that covers general information about alcohol, its effect on the brain and the body, potential risks and harms of drinking, and an account of the threshold values of sensible drinking
  Arms: Usual care
Behavioral: Online multi session follow-up — An online multi session follow-up program (i.e., "Balance"). The central concept of Balance is to support continued self-regulation throughout the behavior change process. There are four key aspects of the program, the first is focus on goal setting and tracking of alcohol consumption on a day-to-day basis. The second on relapse prevention - for example, when clients report drinking more than their target, they receive individualized content aimed at preventing a full blown relapse. The third is emotion regulation, where content and assignments from positive psychology and from cognitive behavioral therapy are used. Finally, intervention covers alcohol education (i.e. the same topics as in the booklet provided to the control group).
  Arms: Extended follow-up

SUMMARY:
The purpose of this study is to test - in a workplace setting - if an online multi-session alcohol intervention improves treatment effect over and above a single session screening with feedback.

Hypothesis: automated online multi-session follow-up improves the effect on alcohol consumption over and above a single session screening

DETAILED DESCRIPTION:
Setting: Online study among Norwegian employees.

Participants: At-risk drinkers among employees in a select group of norwegian workplaces is recruited through an e-mail to their job e-mail account, and advertisements on the intranet of their organization.

Design: Randomized controlled trial (RCT). Subjects in both conditions receives a single session screening procedure including individualized normative feedback. The control group receives an online booklet about the effects of alcohol. The treatment group receives the multi session follow up program "Balance".

ELIGIBILITY:
Inclusion Criteria:

* hazardous or harmful drinking (i.e., a FAST-score of 3 or more)

Exclusion Criteria:

* underage (<18)
* not provided a valid e-mail address
* not provided a valid (Norwegian) mobile phone number

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2011-04; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
The number of standard alcohol units consumed during the previous seven days | Measured six months after enrollment/baseline
  Subjects are asked to indicate (through online questionnaires) how many standard alcohol units they consumed on each of the previous seven days, on a scale from zero to ten. Then a sum-score for weekly consumption is calculated, ranging from zero to 70.

SECONDARY OUTCOMES:
Sick leave during last week | Assessed at six months post baseline
  Sick leave was assessed with a "yes" or "no" response for each of the past seven days, and then accumulated, resulting in a score of zero to seven. Participants were instructed to report any sick leave regardless of reason.
Negative consequences of alcohol consumption | Assessed at six months post baseline
  Perceived negative consequences of own alcohol consumption, during the seven previous days, was assessed by a 13 item index, resulting in a sum score with a theoretical range from zero to 13. The items comprised: headache, nausea, anxiety, worn out, depressed, breaking a plan, breaking a date, sick leave, memory problems, bad conscience, conflict, destroyed something and injuries.

CONTACTS AND LOCATIONS:
Overall Officials: Håvar Brendryen, PhD, Principal Investigator — The Norwegian Centre for Addiction Research, University of Oslo
Locations (1):
- The Norwegian Centre for Addiction Research, University of Oslo, Oslo, Norway

REFERENCES:
- [Background] Brendryen H, Johansen A, Nesvag S, Kok G, Duckert F. Constructing a Theory- and Evidence-Based Treatment Rationale for Complex eHealth Interventions: Development of an Online Alcohol Intervention Using an Intervention Mapping Approach. JMIR Res Protoc. 2013 Jan 23;2(1):e6. doi: 10.2196/resprot.2371. PMID 23612478
- [Derived] Brendryen H, Johansen A, Duckert F, Nesvag S. A Pilot Randomized Controlled Trial of an Internet-Based Alcohol Intervention in a Workplace Setting. Int J Behav Med. 2017 Oct;24(5):768-777. doi: 10.1007/s12529-017-9665-0. PMID 28755326
- See also: The detailed treatment rationale and description of intervention used in the current trial — http://www.researchprotocols.org/2013/1/e6/